CLINICAL TRIAL: NCT06811012
Title: Phase II Clinical Study of Contezolid for the Treatment of Bone and Joint Tuberculosis
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Nie WenJuan, chief physician, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCP-TB-2024-1-31
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis; Bone; Joint
Keywords: Contezolid; tuberculosis; bone; joint
MeSH Terms: conditions — Tuberculosis | interventions — contezolid; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contezolid (Experimental): Contezolid 800mg QD for 14 days
  Interventions: Drug: Contezolid
- linezolid (Active Comparator): Linezolid 600mg QD for 14 days.
  Interventions: Drug: Linezolid (LZD)

INTERVENTIONS:
Drug: Contezolid — This study intends to enroll 24 patients with bone and joint tuberculosis, who will be randomly divided into two groups: the contezolid monotherapy group and the linezolid monotherapy group. Patients will receive oral contezolid or linezolid monotherapy for 14 consecutive days, and data on treatment safety, pharmacokinetics, and preliminary efficacy will be collected before and after administration.
  Study Medications:
  Contezolid 800mg QD for 14 days; Linezolid 600mg QD for 14 days.
  Arms: Contezolid
Drug: Linezolid (LZD) — Linezolid 600mg QD for 14 days.
  Arms: linezolid

SUMMARY:
Contezolid is a novel oxazolidinone antibacterial agent that has shown promising application prospects in the field of tuberculosis treatment in recent years. Studies have demonstrated that contezolid exhibits comparable anti-tuberculosis activity to linezolid both in vitro and in vivo, and even superior intracellular bactericidal activity against Mycobacterium tuberculosis. More importantly, contezolid significantly reduces the risks of bone marrow suppression toxicity, neurotoxicity, and lactic acidosis compared to linezolid, thereby enhancing the drug's safety and tolerability.

In the treatment of bone and joint tuberculosis, contezolid, as a new anti-tuberculosis drug, holds potential significant value. Firstly, it can provide new options for the treatment of drug-resistant Mycobacterium tuberculosis, improving treatment outcomes. Secondly, its lower toxic and side effects can enhance patient compliance, ensuring the smooth progress of treatment. Additionally, contezolid may exhibit synergistic effects with other anti-tuberculosis drugs, further optimizing treatment regimens. Therefore, conducting research on the application of contezolid in the treatment of bone and joint tuberculosis not only helps to improve the cure rate of the disease but also may open up new avenues for the treatment of tuberculosis.

The aim of this study is to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of contezolid in the treatment of bone and joint tuberculosis.

DETAILED DESCRIPTION:
Contezolid is a novel oxazolidinone antibacterial agent that has shown promising application prospects in the field of tuberculosis treatment in recent years. Studies have demonstrated that contezolid exhibits comparable anti-tuberculosis activity to linezolid both in vitro and in vivo, and even superior intracellular bactericidal activity against Mycobacterium tuberculosis. More importantly, contezolid significantly reduces the risks of bone marrow suppression toxicity, neurotoxicity, and lactic acidosis compared to linezolid, thereby enhancing the drug's safety and tolerability.

In the treatment of bone and joint tuberculosis, contezolid, as a new anti-tuberculosis drug, holds potential significant value. Firstly, it can provide new options for the treatment of drug-resistant Mycobacterium tuberculosis, improving treatment outcomes. Secondly, its lower toxic and side effects can enhance patient compliance, ensuring the smooth progress of treatment. Additionally, contezolid may exhibit synergistic effects with other anti-tuberculosis drugs, further optimizing treatment regimens. Therefore, conducting research on the application of contezolid in the treatment of bone and joint tuberculosis not only helps to improve the cure rate of the disease but also may open up new avenues for the treatment of tuberculosis.

The aim of this study is to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of contezolid in the treatment of bone and joint tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* (1) Inpatients who have been diagnosed or clinically diagnosed with bone and joint tuberculosis within the past 3 months prior to screening; (2) Voluntarily participate in this study and sign the informed consent form; (3) Male and female participants must use effective contraception during the study and for 1 month after the study ends.

Exclusion Criteria:

* (1) Patients who have been on long-term corticosteroid therapy or taking immunosuppressants within 90 days prior to screening; (2) Pregnant women, postpartum women, and lactating women; (3) Patients with a history of allergy or known hypersensitivity to contezolid or linezolid, or a history of severe adverse reactions; (4) Evidence of resistance to contezolid or linezolid; (5) Patients deemed unsuitable for participation in this study by the investigator's assessment; (6) Patients whom the investigator believes participation in this study would harm their health, or who are deemed unable to comply with the scheduled visits and assessments as outlined in the protocol, and therefore unsuitable for participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
concentration tests will be conducted on both blood and lesion tissue samples. | 14 days
  After 14 days of oral treatment with contezolid or linezolid, patients will undergo surgery or puncture to obtain tissue from the site of the bone and joint tuberculosis lesion, and concentration tests will be conducted on both blood and lesion tissue samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chest hospital affiliated to Capital medical university, Beijing Tuberculosis & Thoracic Tumor Research Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
In our institution, it is not allowed to post hospital information and patient information on websites for public disclosure.